CLINICAL TRIAL: NCT07154498
Title: Effectiveness of Conventional Physiotherapy Interventions With and Without Cognitive Behavior Therapy on Pain and Quality of Life in Fibromyalgia Patient
Brief Title: Effectiveness of CPI With and Without Cognitive BT on Pain QOL in Fibromyalgia Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/753
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy with Cognitive Behavior Therapy (Experimental)
  Interventions: Behavioral: Conventional physiotherapy with Cognitive Behavior Therapy
- Conventional physiotherapy (Active Comparator)
  Interventions: Combination Product: Conventional physiotherapy

INTERVENTIONS:
Behavioral: Conventional physiotherapy with Cognitive Behavior Therapy — Gentle exercises include stretching and strengthening exercises. Cognitive-behavioral therapy (CBT) sessions.
  Arms: Conventional physiotherapy with Cognitive Behavior Therapy
Combination Product: Conventional physiotherapy — Gentle exercises include stretching and strengthening exercises mobilisation, soft tissue mobilisation Interventions was applied at two sessions per week, each session is about an hour total of 24 sessions. Assessment was done at baseline in the 6th week and 12th week.
  Arms: Conventional physiotherapy

SUMMARY:
The study is a randomized clinical trial conducted at Maryam Hospital Burewala, focusing on the treatment of fibromyalgia in adults aged 18 to 65 years. The sample size was 60+6=66, divided into two groups. The selection criteria included patients with confirmed fibromyalgia diagnosis, persistent symptoms for at least 6 months, and willingness to provide informed consent. Exclusion criteria included other chronic pain conditions, severe psychiatric disorders, substance abuse, unstable medical conditions, or participation in another clinical trial.

DETAILED DESCRIPTION:
The Fibromyalgia Impact Questionnaire (FIQ) and the SF-36 questionnaire were used to assess pain intensity, fatigue, sleep quality, and other symptoms. Subjects were divided into two groups and treated with two sessions per week, each lasting about an hour. The study is single-blind, with assessors and physical therapists being aware of the treatment given to both groups. Data analysis will be performed using SPSS version 24, with normality assessed using the Kolmogorov-Smirnov test. A P-value of ≤ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Confirmed diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) 2010/2011 criteria.
* Adults aged 18 to 65 years.
* Both genders was included
* Persistent symptoms of fibromyalgia for at least 6 months.
* Ability and willingness to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Presence of other chronic pain conditions that could interfere with the assessment of fibromyalgia symptoms (e.g., rheumatoid arthritis, lupus).
* Diagnosis of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder) that could impact the ability to participate in the study.
* Current substance abuse or dependence within the past 6 months
* Presence of unstable or severe medical conditions (e.g., uncontrolled diabetes, severe cardiovascular disease) that could affect participation or pose a risk during the study.
* Participation in another clinical trial within the past 30 days.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire (FIQ) | 12 Months
  The Fibromyalgia Impact Questionnaire (FIQ) is a 10-item, self-administered tool assessing fibromyalgia's impact on physical function, job difficulty, pain, fatigue, and well-being, with a total score from 0 to 100, where higher scores indicate greater impact. The original FIQ uses a 4-point Likert scale for physical function, a 7-day scale for work/feel well days, and visual analog scales (0-10cm) for pain, fatigue, stiffness, anxiety, and depression. Scoring involves normalizing each section and summing them, with specific multipliers and potential adjustments for missing items to reach a total of 100
The Short Form-36 (SF-36) | 12 Months
  The Short Form-36 (SF-36) is a 36-question, patient-reported health survey that measures self-reported health-related quality of life (HRQOL) by assessing eight health domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Responses are scored on a 0-100 scale, where 0 represents maximum disability and 100 represents no disability

CONTACTS AND LOCATIONS:
Locations (1):
- Maryam Hospital Burewala, Burewala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No